CLINICAL TRIAL: NCT01196403
Title: Bladder Cancer: Open Versus Laparoscopic or Robotic Cystectomy. A Study to Determine the Feasibility of Randomization to Open Versus Minimal Access Cystectomy in Patients With Bladder Cancer.
Brief Title: Standard Surgery or Minimal-Access Surgery in Treating Patients With Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000684060; WCTU-BOLERO; ISRCTN-38528926; EU-21069; CRUK-08/036; WCTU-SPON-568-08
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2010-09

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment
Procedure: robot-assisted laparoscopic surgery
Procedure: therapeutic conventional surgery
Procedure: therapeutic laparoscopic surgery

SUMMARY:
RATIONALE: Minimal-access surgery uses a smaller opening in the body to remove the tumor than is used in standard surgery. It is not yet known whether minimal-access surgery to remove the bladder is more effective than standard surgery to remove the bladder in treating patients with bladder cancer.

PURPOSE: This randomized phase II trial is studying standard surgery to see how well it works compared with minimal-access surgery in treating patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of randomizing patients with bladder cancer to undergo an open cystectomy versus a minimal-access cystectomy (laparoscopic or robotic cystectomy).

Secondary

* To assess the safety and efficacy of laparoscopic or robotic cystectomy and the reasons for non-acceptance of randomization.
* To collect safety and toxicity data, including measures of postoperative morbidity and surgical complications. (Exploratory)
* To investigate anatomical lymph node dissection (an indicator for oncological clearance) and completeness of cancer surgery. (Exploratory)
* To determine the quality of life of these patients using EORTC QLQ-C30 and EORTC QLQ-BLM30 questionnaires. (Exploratory)

OUTLINE: This is a multicenter study. Patients who consent to the interview-only (but not randomization) undergo a qualitative interview exploring factors relating to this decision. Patients who consent to randomization are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo an open radical cystectomy.
* Arm II: Patients undergo a minimal-access radical cystectomy (laparoscopic or robotic).

Patients complete quality-of-life questionnaires (EORTC QLQ-C30 and EORTC QLQ-BLM30) at baseline and at 4 weeks, 6 weeks, 8 weeks, 3 months, and 6 months after completion of study therapy. Blood, urine, and tissue samples are collected from some patients at baseline and during study for laboratory analysis.

After completion of study treatment, patients are followed up at 6 weeks, 3 months, and 6 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: A total of 92 patients (72 patients for the randomized portion and 20 for the interview-only portion) are accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed bladder cancer, including any of the following cell types:

  * Urothelial cell (transitional cell) carcinoma
  * Squamous cell carcinoma
  * Adenocarcinoma
* Stage pT1, pT2, or pT3 disease OR mobile bladder mass on bimanual examination under anesthesia
* No enlarged nodes or distant metastases on CT or MRI scan of the abdomen and pelvis
* No upper urinary tract disease

PATIENT CHARACTERISTICS:

* American Society of Anesthesiologist (ASA) status 1-3
* Life expectancy > 24 months
* Not pregnant or nursing
* Negative pregnancy test
* No concurrent disease that would render the patient unsuitable for the trial
* No presence of urosepsis

PRIOR CONCURRENT THERAPY:

* May have received prior neoadjuvant chemotherapy provided study surgery is performed between 3 and 10 weeks from the date of the completion of chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who consent to be randomized

SECONDARY OUTCOMES:
Potential barriers to randomization via semistructured qualitative interviews with patients who consent to registration and do not accept randomization
Potential factors relating to non-registration of patients who are eligible for inclusion but have not been registered based on review of anonymous screening logs
Safety and efficacy
Quality of life data measuring return to normal activities (physical, social, and occupational)

CONTACTS AND LOCATIONS:
Overall Officials: John Kelly, MD, Principal Investigator — University College London Hospitals
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge, England
  - Guy's Hospital, London, England
  - University College of London Hospitals, London, England
  - Wales Cancer Trials Unit, Cardiff, Wales